CLINICAL TRIAL: NCT07281417
Title: Neoadjuvant Chemotherapy With or Without Cemiplimab (REGN2810) in Sinonasal Squamous Cell Carcinoma: A Randomized Phase 2 Study
Brief Title: Testing the Addition of Cemiplimab (REGN2810) to Chemotherapy Treatment Given Prior to Surgery in Patients With Sinonasal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-09016; NCI-2025-09016 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10721 (Other: Ohio State University Comprehensive Cancer Center LAO); 10721 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2025-12-12; First posted 2025-12-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Sinonasal Squamous Cell Carcinoma; Stage III Sinonasal Cancer AJCC v8; Stage IVA Sinonasal Cancer AJCC v8; Stage IVB Sinonasal Cancer AJCC v8
MeSH Terms: interventions — Biopsy; Specimen Handling; Carboplatin; cemiplimab; Chemoradiotherapy; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; Radiotherapy; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (cemiplimab, carboplatin, paclitaxel) (Experimental): See Detailed Description.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Carboplatin; Biological: Cemiplimab; Other: Chemoradiotherapy; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Procedure: Surgical Procedure
- Arm 2 (carboplatin, paclitaxel) (Active Comparator): See Detailed Description.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Carboplatin; Other: Chemoradiotherapy; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Carboplatin — Given carboplatin
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN 2810; REGN-2810; REGN2810
  Arms: Arm 1 (cemiplimab, carboplatin, paclitaxel)
Other: Chemoradiotherapy — Undergo SOC CRT
  Other Names: Chemoradiation; CRT; CRTx; Radiochemotherapy; RCTx; RT-CT
Drug: Cisplatin — Given cisplatin
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo PET/CT and CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase II trial compares the effect of chemotherapy (carboplatin and paclitaxel) with versus without cemiplimab given before surgery (neoadjuvant) in patients with sinonasal squamous cell cancer. Carboplatin is in a class of medications known as platinum-containing compounds. Carboplatin works by killing, stopping or slowing the growth of cancer cells. Paclitaxel is in a class of medications called antimicrotubule agents. It stops cancer cells from growing and dividing and may kill them. Immunotherapy with monoclonal antibodies, such as cemiplimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The usual approach for patients with sinonasal squamous cell cancer is surgery followed by radiation therapy, with or without chemotherapy. Recently, some patients have also been treated with neoadjuvant chemotherapy before surgery. Adding cemiplimab to chemotherapy before surgery may be more effective at stopping the cancer from growing or spreading, compared to chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess whether neoadjuvant therapy (NAT) with cemiplimab (REGN2810)/carboplatin/paclitaxel (Arm 1) results in improved event free survival (EFS) compared to carboplatin/paclitaxel (Arm 2) in participants with sinonasal squamous cell carcinoma (SNSCC).

SECONDARY OBJECTIVES:

I. To compare objective response rate (ORR) between neoadjuvant cemiplimab (REGN2810)/carboplatin/paclitaxel (Arm 1) and neoadjuvant carboplatin/paclitaxel (Arm 2) and to historical standard of care (SOC) in participants with SNSCC.

II. To compare overall survival (OS) between neoadjuvant cemiplimab (REGN2810)/carboplatin/paclitaxel (Arm 1) and carboplatin/paclitaxel (Arm 2) and to historical SOC in participants with SNSCC.

III. To characterize toxicity with NAT in SNSCC. IV. To measure changes in T-cell clonality/diversity using ribonucleic acid (RNA) sequencing (RNAseq) and correlate with NAT response and EFS.

V. To evaluate organ preservation (orbital and skull base) rate with NAT in SNSCC.

CORRELATIVE OBJECTIVES:

I. To correlate human papillomavirus (HPV) status with ORR and OS after NAT. II. To correlate combined positive score (CPS) for PD-L1 expression with OS and EFS.

III. To measure the kinetics of circulating tumor DNA (ctDNA) pre- and post-NAT and correlate with ORR and OS after NAT.

IV. To conduct DNA sequencing on pre-treatment tumor biopsies to determine whether features of the tumor genomic landscape are associated with response to NAT.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1:

NAT: Patients receive cemiplimab intravenously (IV) over 30 minutes on day 1 of each cycle, carboplatin IV over 30 minutes on day 1 of each cycle, and paclitaxel IV over 180 minutes on day 1 of each cycle. Cycles repeat every 21 days (3 weeks) for up to 2 cycles (6 weeks) in the absence of disease progression or unacceptable toxicity. At the discretion of the investigator, patients may alternatively receive carboplatin IV over 30 minutes and paclitaxel IV over 60 minutes weekly during the 2, 3-week cycles. Up to 14 days after completion of NAT, patients are evaluated for response and proceed to definitive therapy.

DEFINITIVE THERAPY: Patients with complete response (CR) or partial response (PR) receive concurrent SOC chemoradiotherapy (CRT). Patients with stable disease (SD) or progressive disease (PD) undergo surgery within 6 weeks of completion of NAT followed by SOC adjuvant therapy.

ADJUVANT THERAPY: Within 4-6 weeks of surgery, patients undergo radiation therapy (RT) once daily, 5 days per week for a total of 30 fractions over 6 weeks and receive cisplatin or carboplatin weekly during RT.

Patients also undergo magnetic resonance imaging (MRI), positron emission tomography (PET)/computed tomography (CT), CT, and collection of blood samples throughout the trial. Patients may undergo biopsy pre-treatment and/or on study.

ARM 2:

NAT: Patients receive carboplatin IV over 30 minutes on day 1 of each cycle and paclitaxel IV over 180 minutes on day 1 of each cycle. Cycles repeat every 21 days (3 weeks) for up to 2 cycles (6 weeks) in the absence of disease progression or unacceptable toxicity. At the discretion of the investigator, patients may alternatively receive carboplatin IV over 30 minutes and paclitaxel IV over 60 minutes weekly during the 2, 3-week cycles. Up to 14 days after completion of NAT, patients are evaluated for response and proceed to definitive therapy.

DEFINITIVE THERAPY: Patients with CR or PR receive concurrent SOC CRT. Patients with SD or PD undergo surgery within 6 weeks of completion of NAT followed by SOC adjuvant therapy.

ADJUVANT THERAPY: Within 4-6 weeks of surgery, patients undergo RT once daily, 5 days per week for a total of 30 fractions over 6 weeks and receive cisplatin or carboplatin weekly during RT.

Patients also undergo MRI, PET/CT, CT, and collection of blood samples throughout the trial. Patients may undergo biopsy pre-treatment and/or on study.

After completion of definitive therapy, patients are followed up at 3, 9, 15, 21, and 27 months and then every 12 months for an additional 3 years (5 years total follow up).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed squamous cell carcinoma of sinonasal origin
* Patients must have a T stage (T3, T4a, and select T4b) primary tumor according to American Joint Committee on Cancer (AJCC) 8th edition. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm (≥ 2 cm) by chest x-ray or as ≥ 10 mm (≥ 1 cm) with CT scan, MRI, or calipers by clinical exam
* No evidence of metastatic disease determined by pre-treatment imaging. Metastatic disease to neck nodes is considered locally advanced and therefore allowable. Patients with N0 and N1-3 disease will be eligible
* Known HPV status (i.e., HPV negative, p16 immunohistochemistry [IHC] positive, high risk [HR]-HPV in situ hybridization [ISH] positive) from testing performed prior to referral. HPV status data (e.g., date of test, type of test [p16 IHC or HR-HPV ISH] and testing result) must be collected during enrollment. Patients who do not have this information available for collection will not be enrolled on this study
* Age ≥ 18 years

  * Because no dosing or adverse event data are currently available on the use of cemiplimab (REGN2810) in combination with carboplatin and paclitaxel in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Hemoglobin ≥ 8 g/dL (acceptable to reach via transfusion)
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 × institutional ULN
* Creatinine clearance ≥ 40 mL/min
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Based on its mechanism of action, cemiplimab (REGN2810) can cause fetal harm when administered to a pregnant woman. Animal studies have demonstrated that inhibition of the PD-1/PD-L1 pathway can lead to increased risk of immune-mediated rejection of the developing fetus resulting in fetal death. For this reason and because paclitaxel is a class D agent with the potential for teratogenic or abortifacient effects, women of childbearing potential (WCBP) and men should use highly effective contraception during treatment and for 6 months after the last dose of the study drugs. WCBP and men should avoid donating eggs/sperm during treatment and for 6 months after the last dose of the study drugs. Women should discontinue nursing during treatment and for 6 months after the last dose of the study drugs
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients with unresectable disease
* Patients presenting with T3 disease without the need for maxillectomy and/or orbital invasion requiring orbital dissection/resection
* Patients who have had any previous systemic therapy to the index lesion in the past 12 months. This includes cemiplimab (REGN2810) and/or other immune modulating agents. Previous systemic therapy may alter or affect response
* Patients who had palliative RT (< 20 Gy) within 1 week prior to entering the study
* Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-mediated adverse events (imAEs)
* History of pneumonitis within the last 5 years
* Patients who have not recovered from adverse events (AEs) due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cemiplimab (REGN2810) or carboplatin and paclitaxel
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because of the increased risk of immune-mediated rejection of the developing fetus with cemiplimab (REGN2810). Men and WCBP who are not prepared to use highly effective contraception during and for 6 months after completion of treatment are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2033-10-03 (Estimated); Study Completion 2033-10-03 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | From randomization to first occurrence of progression of disease or death, assessed up to 5 years
  Progression will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1. To evaluate EFS, survival functions will be computed using the Kaplan-Meier method and compared between groups using the stratified log-rank test. Adjustment for additional covariates will be performed using Cox proportional hazards regression analysis if numbers allow.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 5 years
  ORR will be defined as complete response + partial response (≥ 30% decrease in tumor volume) per Response Evaluation Criteria in Solid Tumors version 1.1 criteria. ORR will be estimated with a 95% confidence interval using the exact Clopper Pearson method. The ORR will be compared between with neoadjuvant cemiplimab (REGN2810)/carboplatin/paclitaxel (Arm 1) to carboplatin/paclitaxel (Arm 2) using the Cochran-Mantel-Haenszel test, stratified by the same factors used for the primary endpoint. ORR for the aggregate study cohort (Arm 1 + Arm 2) will be compared to historical standard of care using the same analysis plan.
Incidence of adverse events (AEs) associated with neoadjuvant therapy (NAT) | Up to 5 years
  Both acute toxicities and chronic toxicities will be graded by the treating investigator using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The frequency of participants experiencing a specific AE will be tabulated by dose level, cycle, seriousness, worst severity, timing of occurrence, outcome, and relationship to study drug. In addition, the number and percentage of participants experiencing a specific toxicity will be tabulated similarly. Accrual will be halted if excessive numbers of unacceptable toxicities are observed. This is defined as > 30% grade 4 treatment-related AEs, which are directly attributable to NAT.
Changes in T-cell clonality/diversity | Up to 5 years
  The changes in T-cell clonality/diversity will be assessed using ribonucleic acid sequencing (RNAseq) and correlated with NAT response and EFS. RNAseq data will undergo quality control, alignment to the human reference genome, and transcript quantification using standard bioinformatics pipelines. T-cell receptor sequences will be reconstructed using tools such as MiXCR or TRUST4. Measures of T-cell clonality and diversity (e.g., Shannon entropy, clonality index) will be calculated. Changes in T-cell clonality/diversity pre- and post-treatment will be assessed using paired t-tests or Wilcoxon signed-rank tests. Associations with NAT response and EFS will be analyzed using logistic regression and Cox proportional hazards models, adjusting for relevant covariates. Multiple testing correction using the Benjamini-Hochberg method will be applied where appropriate.
Organ preservation rates | Up to 5 years
  Organ preservation in the post-treatment setting is defined as physical and functional preservation of the organ. For example, orbital preservation would imply maintenance of the entirety of the orbit and preservation of vision and motion. Orbital preservation rates will be summarized using descriptive statistics such as mean, standard deviation, median, and range. At the time of enrollment the treating team, with the guidance of the surgical team, will indicate what major anatomic locations would have to be resected if the patient elected initial primary surgical therapy (palate, orbit, and/or skull base). This prospective information will allow concrete subsequent secondary analyses of organ preservation rates without the bias of outcome or recall.
Overall survival (OS) | From the start of NAT to death, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate OS and 95% confidence intervals will be reported. OS for the aggregate study cohort (Arm 1 + Arm 2) will be compared to historical standard of care using the same analysis plan.

OTHER OUTCOMES:
OS | From the start of NAT to death, assessed up to 5 years
  Will correlate human papillomavirus status, combined positive score for PD-L1 expression, and circulating tumor deoxyribonucleic acid (ctDNA) with OS.
EFS | From randomization to first occurrence of progression of disease or death, assessed up to 5 years
  Will correlate human papillomavirus status, combined positive score for PD-L1 expression, and ctDNA with EFS.
NAT response rates | Up to 5 years
  Will correlate human papillomavirus status, combined positive score for PD-L1 expression, and ctDNA with NAT response rates.
ctDNA | At pre-treatment, in weeks 7-8 (post-NAT visit), and at 3 months following definitive treatment
  ctDNA will be measured at pre-defined timepoints. Sequencing using whole exome sequencing will be conducted on pre-treatment tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Sheth, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm